CLINICAL TRIAL: NCT02198417
Title: Effects of Metformin on Mitochondrial Function in Polycystic Ovary Syndrome
Brief Title: Metformin Treatment in Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Utah (Other)
Responsible Party: Principal Investigator, Corrine Welt, Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014P000911; R01HD065029 (NIH)
Record Dates: First submitted 2014-07-17; First posted 2014-07-23 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; PCOS; Acne; Infertility; Irregular menses; Irregular period; Mitochondria; Metabolism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Acne Vulgaris; Infertility; Menstruation Disturbances | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental): Metformin ER 1500 mg per day treatment for 12 weeks
  Interventions: Drug: Metformin ER

INTERVENTIONS:
Drug: Metformin ER — Treatment with metformin ER for 12 weeks
  Other Names: Glucophage

SUMMARY:
PCOS occurs when a woman does not release an egg regularly each month, causing her periods to be irregular. Women with PCOS can also have increased hair growth on the face and body, acne, head balding, infertility, pre-diabetes, and diabetes. PCOS is commonly treated with oral contraceptive pills (also known as the birth control pills). Sometimes, a medication called metformin is also used to treat PCOS, especially if a woman has evidence of insulin resistance or if fertility is desired. Unfortunately, metformin works in only some women with PCOS. The mechanism through which metformin works in PCOS is not clear and it difficult to predict who will benefit from metformin treatment and who will not.

The investigators are doing this research study to look at how the medication metformin affects the cells in the body of patients with PCOS. Specifically, the investigators will look at how metformin affects the mitochondria. Mitochondria are the part of cells that produce fuel (energy) for other cells and play a role in metabolism. The investigators would like to see whether there is a relationship between mitochondrial activity and symptoms of polycystic ovary syndrome (PCOS) before and after treatment with metformin. They would also like to study whether genes affect the response to metformin in women with PCOS.

DETAILED DESCRIPTION:
Women who are eligible to enroll in this study will be treated with the medication metformin for 12 weeks. Before and after treatment with metformin, the following will be assessed:

* Weight, blood pressure, waist circumference
* Lipids (cholesterol)
* Hormone levels (including testosterone and other androgens)
* IV glucose tolerance test (to assess for early evidence of insulin resistance)
* Effect of metformin on muscle mitochondria (this will involve one MRI scan and one muscle biopsy each before and after treatment with metformin)

Ovulation will be closely monitored at least twice a month with pelvic ultrasounds and blood tests for estrogen and progesterone levels.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome
* No hormonal or antidiabetic medications for 1 month
* Good general health

Exclusion Criteria:

* Smoker
* Acute infection or chronic disease
* Diabetes
* Pregnant or trying to get pregnant over next half year
* Bleeding disorders
* Any metal or foreign implants (e.g., aneurysm clips, ear implants, heart pacemakers or defibrillators)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Muscle Metabolism/Mitochondrial Function | 3 months
  The change in mitochondrial activity before and after metformin treatment will be analyzed in relationship to the clinical response to 3 months of metformin treatment (i.e., clinical response to metformin = changes in glucose metabolism, hormone levels, and ovulation response)

SECONDARY OUTCOMES:
Genetic risk variants affecting mitochondrial function/metabolism | 3 months
  Blood will be analyzed for differences in genes between patients and its relationship to mitochondrial function.

CONTACTS AND LOCATIONS:
Overall Officials: Corrine Welt, M.D., Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Background] Pau CT, Keefe C, Duran J, Welt CK. Metformin improves glucose effectiveness, not insulin sensitivity: predicting treatment response in women with polycystic ovary syndrome in an open-label, interventional study. J Clin Endocrinol Metab. 2014 May;99(5):1870-8. doi: 10.1210/jc.2013-4021. Epub 2014 Feb 25. PMID 24606093